CLINICAL TRIAL: NCT06237569
Title: Effects of Low Dose ketamıne on Postpartum Depression During Caesarean Sections
Brief Title: Dose Low Dose Ketamine in Casesarian
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DUYGU DEMİROZ, principal investigator, Inonu University
Other Study IDs: inonu Caesarean
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain; Postpartum Depression
Keywords: midazolam with low dose ketamine; low dose ketamine; postoperatıve analgesıc need; postpartum depression
MeSH Terms: conditions — Pain, Postoperative; Depression, Postpartum | interventions — Midazolam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Grup 1 -Ketamine Group: Ketamine Group (GROUP 1) 0.5 mg/kg IV single dose bolus diluted to 5 ml with 0.9% saline
  Interventions: Drug: Application of ketamine and midazolam or ketamine alone to patients undergoing cesarean section under spinal anesthesia
- Group 2-ketamine + midazolam: Midazolam 0.0125 mg/kg is given followed by a single IV bolus dose of 0.5 mg/kg diluted to 5 ml with 0.9% saline.
  Interventions: Drug: Application of ketamine and midazolam or ketamine alone to patients undergoing cesarean section under spinal anesthesia
- Group 3-placebo: Group 3-placebo ;A single dose of IV 5 ml physiological saline will be given.
  Interventions: Drug: Application of ketamine and midazolam or ketamine alone to patients undergoing cesarean section under spinal anesthesia

INTERVENTIONS:
Drug: Application of ketamine and midazolam or ketamine alone to patients undergoing cesarean section under spinal anesthesia — A single dose of 0.5 mg/kg IV diluted to 5 ml with 0.9% saline was planned to be administered simultaneously to the Ketamine Group (GROUP 1), ketamine and midazolam within 5 minutes after the newborn umbilical cord was clamped (Group 2). After midazolam 0.03 mg/kg is given, a single dose IV bolus of 0.5 mg/kg diluted to 5 ml with 0.9% saline will be administered.
  Patients experience dizziness, hallucinations, nausea, headache, vomiting, diplopia and blurred vision, the time until the first analgesic request; Depression parameters will be evaluated with the Edinburgh Postpartum Depression Scale (EPDS) in all patients before cesarean section and at the 1st, 2nd and 4th weeks after birth.

SUMMARY:
The results of ketamine, ketamine and midazolom and placebo can be copied after birth in cesareans subjected to spinal anesthesia.

DETAILED DESCRIPTION:
Postpartum depression will be evaluated by dividing the patients into 3 groups: group 1 as ketamine, group 2 as ketamine and midasom, and group 3 as placebo group.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists 2-.3 18 -45years old Patients planned to be born by cesarean section The patient requests a cesarean section with spinal anesthesia

ExclusionCriteria:

Pathological obstetric complications

Hypertension

Contraindication for ketamine Contraindication for spinal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — being a patient undergoing cesarean section
Study Population: Patients undergoing cesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
postpartum depression | 4 weeks
  Reducing postpartum depression with low-dose ketamine
intraoperative complications | 1 day
  Reducing postpartum depression by reducing ketamine-related intraoperative complications
postoperative pain | 1 day
  Reducing postoperative pain with low dose ketamine

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU DEMIROZ, Principal Investigator — Inonu University
Locations (1):
- Inonu universitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided